CLINICAL TRIAL: NCT05732545
Title: Application of Enteral Nutrition Program in Patients With Intra-abdominal Hypertension Oriented by Intra-abdominal Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-0899
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Intra-Abdominal Hypertension
Keywords: Intra-Abdominal Hypertention; Enteral Nutrition; Feeding Intolerance
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enteral nutrition program by intra-abdominal pressure (Experimental): enteral nutrition program for patients with intra-abdominal hypertension guided by intra-abdominal pressure
  Interventions: Behavioral: enteral nutrition program for patients with abdominal hypertension guided by abdominal pressure
- Routine nursing measures (No Intervention): Routine nursing measures

INTERVENTIONS:
Behavioral: enteral nutrition program for patients with abdominal hypertension guided by abdominal pressure — There are 4 aspects of intra-abdominal pressure monitoring, source control and treatment for the etiology of increased abdominal pressure, enteral nutrition program, enteral nutrition tolerance evaluation and treatment
  Arms: enteral nutrition program by intra-abdominal pressure

SUMMARY:
In this study, relevant contents of the enteral nutrition nursing programs for severe patients with abdominal pressure were systematically searched, and quality evaluation was carried out based on existing evidence. Based on evidence-based evidence, an enteral nutrition nursing program for patients with abdominal pressure was constructed, to improve the feed tolerance of patients with abdominal pressure, increase nutritional compliance rate, and improve patient prognosis.

DETAILED DESCRIPTION:
Background: Enteral nutrition is the preferred method of artificial nutrition for critically ill patients. Early enteral nutrition within 24 to 48 hours after admission can maintain intestinal mucosal barrier function, increase local blood flow, reduce bacterial migration, and reduce the incidence of intestinal infections. Increased abdominal pressure is considered to be an independent risk factor for feeding intolerance in severe patients. Patients with abdominal pressure are prone to complications such as diarrhea, abdominal distension, vomiting, and even aspiration, which forces the suspension or suspension of enteral nutrition and leads to insufficient nutritional intake in patients. At present, there is evidence that regulating enteral nutrition through monitoring intra-abdominal pressure can effectively reduce the incidence of feeding intolerance in patients. Domestic and foreign scholars have formulated nutrition management programs for patients with intra-abdominal pressure from different aspects, such as monitoring and grading of intra-abdominal pressure, evaluation and management of tolerance, and prevention of complications. However, The standardized enteral nutrition feeding program oriented by the monitoring of intra-abdominal pressure has not yet formed a unified standard.

Objective: This study conducted a quality evaluation based on existing evidence, adopted evidence-based research methods to establish an enteral nutrition program for patients with abdominal hypertension oriented by abdominal pressure, and aimed to improve the feeding tolerance of patients with abdominal hypertension, improve the nutritional compliance rate and improve the prognosis of patients through the implementation of evidence-based practice programs.

ELIGIBILITY:
1. Inclusion Criteria

   1. 12mmHg≤ intraperitoneal pressure ≤20mmHg (1mmHg=0.133kPa)
   2. ≥18 years of age
   3. Consistent with the indications of early enteral nutrition

      * Patients with nutritional risk, gastrointestinal function, or partial gastrointestinal function and unable to eat through the mouth

        * Stable hemodynamics (MAP > 65mmHg, blood lactic acid < 4mmol/L, and vasoactive drugs in the process of reduction or withdrawal)
   4. Patients or their family members sign the informed consent
2. Exclusion Criteria

   1. Pregnant or lactating female patients
   2. Patients with recent abdominal surgery
   3. Patients with a large number of abdominal effusions;
   4. There are contraindications to enteral nutrition

      * Uncontrolled shock

        * Uncontrolled hypoxemia and acidosis

          * Uncontrolled upper gastrointestinal bleeding

            * GRV > 500mL/ 6h

              * Intestinal ischemia

                * Intestinal obstruction

                  * Abdominal space syndrome (ACS)

                    * High fistula without distal feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of feeding intolerance | 7 days
  Incidence of feeding intolerance: refers to the frequency of new cases of feeding intolerance within 7 days after the initiation of enteral nutrition.

SECONDARY OUTCOMES:
The standard rate of feeding | 7 days
  Enteral nutrition feeding standard rate (%)=(actual feeding quantity ÷ target feeding quantity)×100%

CONTACTS AND LOCATIONS:
Locations (1):
- Feng Xiuqin, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No